CLINICAL TRIAL: NCT06560736
Title: Development of Novel Psychological Assessment Tools and Anxiety Intervention for PKU: Intervention Trial
Brief Title: Development of Novel Psychological Assessment Tools and Anxiety Intervention for Phenylketonuria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National PKU Alliance (Unknown)
Responsible Party: Principal Investigator, Shawn Christ, Associate Professor of Psychological Sciences, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2103266
Record Dates: First submitted 2024-04-30; First posted 2024-08-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Wait-list Control Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Other)
  Interventions: Behavioral: Show Me FIRST coping skills intervention
- Wait List / Delayed Intervention Group (Other)
  Interventions: Behavioral: Show Me FIRST coping skills intervention

INTERVENTIONS:
Behavioral: Show Me FIRST coping skills intervention — Show Me FIRST is a flexible, transdiagnostic intervention organized around well-tested principles of youth psychotherapeutic change.

SUMMARY:
While previous PKU intervention research has largely focused on pharmacological treatment of elevated Phe levels, the adaptation of evidence-based psychosocial therapy holds promise for addressing cognitive and psychological symptoms and significantly improving quality of life. Study goals include: (1) to demonstrate the efficacy and feasibility of a short-term skills-based intervention (Show Me FIRST) for anxiety and depression in adolescents with PKU, and (2) to further establish the psychometric validity of novel assessment measures recently developed by the Investigators that utilize ecological momentary assessment (EMA) to capture "in the moment" neurocognitive and psychological function. The Investigators propose to conduct a randomized controlled trial wherein 30 adolescents with PKU will be randomized to either an immediate intervention group or wait-list/delayed intervention group.

DETAILED DESCRIPTION:
A sample of 30 adolescents (age 10-17) with PKU and a history of elevated anxiety and/or depression symptomatology will be recruited to participate in a randomized control trial. Following screening and informed consent, participants will be randomized to an immediate intervention group (n=15) or wait-list/delayed intervention group (n=15). Participants will receive the 10-week Show Me First program for treatment of anxiety and depression. Participants will complete extensive psychological and neurocognitive evaluations at three timepoints: Weeks 0, 11, and 22. The assessments and intervention will all be administered remotely via secure videoconference and cell-phone based applications.

ELIGIBILITY:
Inclusion Criteria:

* Youth 10-17 years old and at least one parent/guardian
* Formal diagnosis of PKU (as confirmed/reported by caregiver): identified by newborn screening with PKU as evidenced by a blood Phe level ≥ 360μmol/L; received treatment within the first 30 days of life.
* Interest in receiving a brief, psychotherapeutic skills program to prevent and treat symptoms of anxiety and/or depression, according to parent- and youth-report
* Located in Missouri, Kansas, or Illinois.

Exclusion Criteria:

* Have significant intellectual disability (IQ<70) or significant expressive or receptive language that would interfere with psychotherapy, according to parent- or youth-report
* Plans to receive non-study psychotherapy during the course of study participation, according to parent- or youth-report
* Plans to change current psychoactive or PKU-related medication during the course of study participation, according to parent- or youth-report
* Have active suicidal ideation that would necessitate immediate treatment or require higher level of care than brief psychotherapy, according to parent- or youth-report

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Anxiety & Depression scales | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of anxiety & depression symptoms
Test My Brain phone-based EMA cognitive test | Weeks 0, 11, & 22
  Performance-based measure of cognitive skill & attention

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of everyday symptoms of executive problems
Blood Phenylalanine Levels | Weeks 0, 5, 11, 16, & 22
ADHD Rating Scale - 4th version (ADHD-RS-IV) | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of ADHD symptoms
Executive Function, Attention, and Speed Symptom Inventory (EASSI) for PKU | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of cognitive symptoms
Rey Auditory Verbal Learning Test (Rey AVLT) | Weeks 0, 11, & 22
  Performance-based measure of memory & learning
Stop Signal Task (SST) | Weeks 0, 11, & 22
  Performance-based measure of inhibitory ability
Revised Children's Anxiety and Depression Scale (RCADS) | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of anxiety & depression symptoms
Behavior & Feelings Survey (BFS) | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of internalizing & externalizing problems
Adolescent Insomnia Questionnaire (AIQ) | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of sleep problems
Global Impression Scale | Weeks 0, 11, & 22
  Patient-reported outcome (PRO) measure of overall symptom severity and improvement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No